CLINICAL TRIAL: NCT00673452
Title: Flexible Dosed Duloxetine Versus Placebo in the Treatment of Fibromyalgia
Brief Title: A Study Comparing Duloxetine and Placebo in the Treatment of Fibromyalgia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12220; F1J-US-HMGB (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2010-06-24 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2010-05

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental): 60-120 mg, oral, every day, 12 weeks
  Interventions: Drug: duloxetine hydrochloride
- Placebo (Placebo Comparator): oral, daily, 12 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: duloxetine hydrochloride — 60-120 mg, oral, every day, 12 weeks (acute blinded phase followed by a 12 week blinded continuation phase).
  Other Names: LY248686; Cymbalta
  Arms: Duloxetine
Drug: placebo — oral, daily, 12 weeks (acute blinded phase followed by 12 weeks of blinded duloxetine treatment)
  Arms: Placebo

SUMMARY:
The purpose of this study is to confirm the efficacy and safety of duloxetine 60-120 mg once daily in comparison to placebo on symptom improvement in patients meeting criteria for fibromyalgia aged 18 and older. Patients will be randomized to duloxetine or placebo, however, all patients will receive duloxetine at some point in the study.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients
* aged 18 and older who meet criteria for fibromyalgia as defined by the American College of Rheumatology
* have a score of at least 4 on the average pain item of the Brief Pain Inventory (BPI) (modified short form) at visits 1 and 2
* all females must test negative for pregnancy at the time of enrollment
* have a degree of understanding such that the patient can provide informed consent, complete protocol required assessments and communicate intelligibly with the investigator and study coordinator.

Exclusion Criteria:

* have pain symptoms related to traumatic injury, structural rheumatic disease, or regional rheumatic disease that will interfere with interpretation of outcome measures
* have regional pain syndrome, multiple surgeries or failed back syndrome
* have confirmed current or previous diagnosis of rheumatoid arthritis, inflammatory arthritis, or infectious arthritis, or an autoimmune disease (i.e. systemic lupus erythematosus)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2008-06; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (46):
- United States (43):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pasadena, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cromwell, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danbury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bradenton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeLand, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oak Brook, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lafayette, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prairie Village, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rockville, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belmont, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fall River, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newton, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edison, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Piscataway, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greensboro, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toledo, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eugene, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Myrtle Beach, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Jackson, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waco, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita Falls, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Jordan, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tacoma, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middleton, Wisconsin
- Puerto Rico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hato Rey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan

REFERENCES:
- [Derived] Mohs R, Mease P, Arnold LM, Wang F, Ahl J, Gaynor PJ, Wohlreich MM. The effect of duloxetine treatment on cognition in patients with fibromyalgia. Psychosom Med. 2012 Jul-Aug;74(6):628-34. doi: 10.1097/PSY.0b013e31825b9855. Epub 2012 Jun 28. PMID 22753629
- [Derived] Arnold LM, Wang F, Ahl J, Gaynor PJ, Wohlreich MM. Improvement in multiple dimensions of fatigue in patients with fibromyalgia treated with duloxetine: secondary analysis of a randomized, placebo-controlled trial. Arthritis Res Ther. 2011 Jun 13;13(3):R86. doi: 10.1186/ar3359. PMID 21668963
- [Derived] Arnold LM, Clauw D, Wang F, Ahl J, Gaynor PJ, Wohlreich MM. Flexible dosed duloxetine in the treatment of fibromyalgia: a randomized, double-blind, placebo-controlled trial. J Rheumatol. 2010 Dec;37(12):2578-86. doi: 10.3899/jrheum.100365. Epub 2010 Sep 15. PMID 20843911
- See also: Lilly Clinical Trials Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients were on duloxetine in the continuation phase. The continuation phase was for exploratory purpose only, and the results will not be presented further.
Groups:
- Duloxetine: 60-120 mg, oral, daily, 12 weeks
Period: Acute Double-Blind Phase
Arm/Group | Duloxetine | Placebo
Started | 263 | 267
Completed | 176 | 187
Not Completed | 87 | 80
Not completed — Adverse Event | 41 | 24
Not completed — Lack of Efficacy | 9 | 14
Not completed — Lost to Follow-up | 16 | 19
Not completed — Physician Decision | 0 | 6
Not completed — Protocol Violation | 5 | 3
Not completed — Sponsor Decision | 0 | 1
Not completed — Withdrawal by Subject | 16 | 13
Period: Continuation Double-Blind Phase
Arm/Group | Duloxetine | Placebo
Started | 176 | 187 (Patients on placebo in acute phase received 60 mg duloxetine during the continuation phase.)
Completed | 151 | 153
Not Completed | 25 | 34
Not completed — Adverse Event | 5 | 13
Not completed — Withdrawal by Subject | 9 | 5
Not completed — Lost to Follow-up | 4 | 5
Not completed — Lack of Efficacy | 2 | 5
Not completed — Protocol Violation | 2 | 3
Not completed — Sponsor Decision | 0 | 3
Not completed — Physician Decision | 2 | 0
Not completed — Death - Cervical vertebral fracture | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 263 | 267 | 530
Age Continuous [Mean (Standard Deviation); unit: years] | 50.74 (11.26) | 49.62 (10.84) | 50.18 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 244 | 250 | 494
  Male | 19 | 17 | 36
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 204 | 206 | 410
  Hispanic | 37 | 46 | 83
  Other - Not Specified | 22 | 15 | 37
Region of Enrollment [Number; unit: participants]
  United States | 263 | 267 | 530
Alcohol Consumption [Number; unit: participants]
  Yes | 89 | 90 | 179
  No | 174 | 177 | 351
Generalized Anxiety Disorder (GAD) Status [Number; unit: participants] — GAD as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV).
  participants
    Yes | 19 | 24 | 43
    No | 244 | 243 | 487
Major Depressive Disorder (MDD) Status [Number; unit: participants] — MDD as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV).
  participants
    Yes | 44 | 53 | 97
    No | 219 | 214 | 433
Tobacco Use [Number; unit: participants]
  Yes | 57 | 42 | 99
  No | 206 | 225 | 431
Beck Anxiety Inventory (BAI) Total Score [Mean (Standard Deviation); unit: units on a scale] — Beck Anxiety Inventory (BAI) is a 21-item patientcompleted questionnaire designed to assess characteristics of anxiety. Each item is rated on a 4-point scale (0 = not present; 3 = present in the extreme). This questionnaire will be used to rate the severity of anxiety symptoms and any improvement during the course of the trial. The total score ranges from 0 to 63; the higher the score, the more severe the anxiety symptoms.
  units on a scale | 12.83 (9.28) | 13.18 (9.77) | 13.00 (9.52)
Beck Depression Inventory II (BDI-II) Total Score [Mean (Standard Deviation); unit: units on a scale] — Beck Depression Inventory-II (BDI-II) is a 21-item patient-completed questionnaire designed to assess characteristics of depression. Each item is rated on a 4-point scale (0 = not present; 3 = present in the extreme). This questionnaire will be used to rate the severity of depressive symptoms and any improvement during the course of the trial. The total score ranges from 0 to 63; the higher the score, the more severe the depressive symptoms.
  units on a scale | 16.16 (10.43) | 16.20 (10.35) | 16.18 (10.38)
Brief Pain Inventory (BPI) Average Pain Score [Mean (Standard Deviation); unit: units on a scale] — A self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
  units on a scale | 6.45 (1.54) | 6.46 (1.62) | 6.45 (1.58)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 163.00 (8.38) | 163.75 (8.48) | 163.38 (8.43)
Likert Scale Rating of Mood, Anxiety, Sleep, Pain, and Stiffness [Mean (Standard Deviation); unit: units on a scale] — Patient-rated likert scale assessment of: Mood - feeling low, sad or depressed (0 = not feeling low, sad or depressed to 10 = feeling extremely low, sad, or depressed); Anxious - anxious feelings (0 = not feeling anxious to 10 = extremely anxious); Sleep - how much patient is bothered by sleep difficulties (0 = not bothered to 10 = extremely bothered); Pain - how much patient is bothered by painful physical discomforts (0 = not bothered to 10 = extremely bothered); Stiffness - how stiff patient has felt in past 24 hours (0 = has not felt any stiffness to 10 = has felt extremely stiff).
  units on a scale
    Anxiety | 3.68 (2.81) | 4.08 (2.90) | 3.88 (2.86)
    Mood | 3.78 (2.76) | 4.04 (2.77) | 3.91 (2.77)
    Pain | 7.25 (1.87) | 7.45 (1.83) | 7.35 (1.85)
    Sleep | 6.74 (2.56) | 6.81 (2.67) | 6.78 (2.62)
    Stiffness | 7.02 (2.00) | 7.12 (1.84) | 7.07 (1.92)
Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (MGH-CPFQ) Total [Mean (Standard Deviation); unit: units on a scale] — The MGH-CPFQ is a self-report instrument consisting of seven questions pertaining to an individual's cognitive and physical well-being. Each question is rated 1 = "greater than normal" to 6 = "totally absent". Total score ranges from 7 to 42.
  units on a scale | 26.71 (6.33) | 26.63 (6.29) | 26.67 (6.30)
Patient's Global Impressions of Severity (PGI-S) [Mean (Standard Deviation); unit: units on a scale] — The PGI-Severity scale is a patient-rated instrument that measures perceived severity of symptoms. It is a 7-point scale where a score of 1 indicates that the patient is "Normal, not at all ill," a score of 4 indicates that the patient has experienced "Moderately ill," and a score of 7 indicates that the patient is "Among the most extremely ill patients."
  units on a scale | 3.88 (1.24) | 3.66 (1.43) | 3.77 (1.34)
The Multidimensional Fatigue Inventory (MFI) Dimension Scores [Mean (Standard Deviation); unit: units on a scale] — The Multidimensional Fatigue Inventory (MFI) is a 20- item, self-reporting instrument designed to collect data on the following 5 dimensions: general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity. Each dimension score is derived by summing the scores of the 4 individual items that pertain to each dimension. Item scores range from 1 to 5; thus, dimensional scores range from 4 to 20 with a higher score reflecting greater levels of fatigue.
  units on a scale
    General Fatigue Dimension | 17.05 (2.91) | 17.16 (2.87) | 17.11 (2.89)
    Mental Fatigue Dimension | 13.28 (4.17) | 12.97 (4.30) | 13.12 (4.24)
    Physical Fatigue Dimension | 15.48 (3.50) | 15.40 (3.61) | 15.44 (3.55)
    Reduced Activity Dimension | 13.78 (4.06) | 13.57 (3.90) | 13.67 (3.98)
    Reduced Motivation Dimension | 12.41 (3.69) | 12.59 (3.70) | 12.50 (3.70)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 84.01 (19.76) | 85.98 (21.65) | 85.00 (20.74)

OUTCOME MEASURES:

1. Primary Outcome: Patient's Global Impressions of Improvement (PGI-I) at Week 12
Description: The PGI-Improvement scale is a patient-rated instrument that measures perceived improvement in symptoms. It is a 7-point scale where a score of 1 indicates that the patient is "very much improved," a score of 4 indicates that the patient has experienced "no change," and a score of 7 indicates that the patient is "very much worse."
Time Frame: 12 weeks
Population: Number of randomized patients with baseline PGI-S and at least one post-baseline PGI-I data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 245 | 255
units on a scale | 2.79 (0.10) | 3.36 (0.09)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Patients treated with 60-120 mg duloxetine for 12 weeks compared with placebo will show greater improvement in symptoms as assessed by Patient's Global Impressions of Improvement (PGI-I). Sample size determined using 2-sided t-test with significance level of 0.05, and discontinuation rate of 5% without postbaseline data. With 261 patients per arm, study has approximately 85% power to detect treatment group difference of -0.4 points (standard deviation of 1.5) in PGI-I between treatment groups; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The a priori threshold for statistical significance was 0.05; Mixed Model Repeated Measures (MMRM) Model: PGI-S = baseline PGI-S + treatment + pooled investigator + visit + treatment-by-visit + baseline-by-visit

2. Secondary Outcome: Change From Baseline in Brief Pain Inventory (BPI) (Modified Short Form) at 12 Week Endpoint
Description: BPI is a self-reported form that assesses severity of pain and the interference of pain on function. There are 4 questions assessing the severity for worst pain, least pain, and average pain in the past 24 hours, and the pain right now. Severity scores range from 0 (no pain) to 10 (pain as bad as you can imagine). There are 7 questions assessing the interference of pain in the past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline, 12 weeks
Population: Number of patients with a non-missing baseline and at least one post-baseline record. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 249 | 258
units on a scale
  Worst Pain Severity | -2.32 (0.17) | -1.57 (0.17)
  Least Pain Severity | -1.57 (0.14) | -0.96 (0.14)
  Average Pain Severity | -2.14 (0.15) | -1.40 (0.15)
  Pain Right Now Severity | -2.10 (0.17) | -1.34 (0.17)
  General Activity Interference | -2.38 (0.17) | -1.44 (0.17)
  Mood Interference | -2.56 (0.18) | -1.61 (0.18)
  Walking Ability Interference | -2.16 (0.17) | -1.36 (0.17)
  Normal Work Interference | -2.37 (0.17) | -1.60 (0.17)
  Relations with Other People Interference | -2.17 (0.17) | -1.22 (0.16)
  Sleep Interference | -2.69 (0.18) | -1.81 (0.18)
  Enjoyment of Life Interference | -2.84 (0.19) | -1.45 (0.19)
  Average Interference | -2.44 (0.16) | -1.52 (0.15)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Worst Pain Severity. P-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: BPI Score change from baseline to LOCF endpoint = BPI baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.75, 95% CI 2-sided [-1.19 to -0.31] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA — P-value for Least Pain Severity. P-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: BPI Score change from baseline to LOCF endpoint = BPI baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.61, 95% CI 2-sided [-0.99 to -0.24] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Average Pain Severity. P-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: BPI Score change from baseline to LOCF endpoint = BPI baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.74, 95% CI 2-sided [-1.13 to -0.35] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Pain Right Now Severity. P-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: BPI Score change from baseline to LOCF endpoint = BPI baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.76, 95% CI 2-sided [-1.20 to -0.31] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for General Activity Interference. P-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: BPI Score change from baseline to LOCF endpoint = BPI baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.94, 95% CI 2-sided [-1.39 to -0.49] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Mood Interference. P-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: BPI Score change from baseline to LOCF endpoint = BPI baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.95, 95% CI 2-sided [-1.41 to -0.49] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Walking Ability Interference. P-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: BPI Score change from baseline to LOCF endpoint = BPI baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.80, 95% CI 2-sided [-1.24 to -0.36] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Normal Work Interference. P-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: BPI Score change from baseline to LOCF endpoint = BPI baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.76, 95% CI 2-sided [-1.21 to -0.32] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 9: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Relations with Other People Interference. P-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: BPI Score change from baseline to LOCF endpoint = BPI baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.95, 95% CI 2-sided [-1.38 to -0.52] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 10: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Sleep Interference. P-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: BPI Score change from baseline to LOCF endpoint = BPI baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.87, 95% CI 2-sided [-1.35 to -0.39] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 11: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Enjoyment of Life Interference. P-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: BPI Score change from baseline to LOCF endpoint = BPI baseline + treatment + pooled investigator; Least Squares Mean Difference = -1.39, 95% CI 2-sided [-1.92 to -0.86] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 12: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Average Interference. P-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: BPI Score change from baseline to LOCF endpoint = BPI baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.93, 95% CI 2-sided [-1.33 to -0.52] — Least Squares Mean Difference = Duloxetine minus Placebo

3. Secondary Outcome: Change From Baseline in Multidimensional Fatigue Inventory (MFI) at 12 Week Endpoint
Description: MFI is a 20-item, self-reporting instrument designed to collect data on the following 5 dimensions: general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity. Each dimension score is derived by summing the scores of the 4 individual items that pertain to each dimension. Item scores range from 1 to 5; thus, dimensional scores range from 4 to 20 with a higher score reflecting greater levels of fatigue.
Time Frame: Baseline, 12 weeks
Population: Number of patients with a non-missing baseline and at least one post-baseline record.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 246 | 254
units on a scale
  General Fatigue | -2.21 (0.22) | -1.38 (0.22)
  Physical Fatigue | -2.08 (0.22) | -1.35 (0.22)
  Mental Fatigue | -2.01 (0.23) | -1.09 (0.23)
  Reduced Activity | -1.46 (0.24) | -0.59 (0.23)
  Reduced Motivation | -1.66 (0.22) | -0.72 (0.21)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.005, ANCOVA — P-value for General Fatigue. P-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.05; Model: MFI subscale change from baseline at endpoint = MFI subscale baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.83, 95% CI 2-sided [-1.41 to -0.25] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.013, ANCOVA — P-value for Physical Fatigue. P-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.05; Model: MFI subscale change from baseline at endpoint = MFI subscale baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.72, 95% CI 2-sided [-1.30 to -0.15] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value for Mental Fatigue. P-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.05; Model: MFI subscale change from baseline at endpoint = MFI subscale baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.92, 95% CI 2-sided [-1.52 to -0.32] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.005, ANCOVA — P-value for Reduced Activity. P-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.05; Model: MFI subscale change from baseline at endpoint = MFI subscale baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.88, 95% CI 2-sided [-1.49 to -0.26] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Reduced Motivation. P-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.05; Model: MFI subscale change from baseline at endpoint = MFI subscale baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.94, 95% CI 2-sided [-1.49 to -0.38] — Least Squares Mean Difference = Duloxetine minus Placebo

4. Secondary Outcome: Change From Baseline in Beck Depression Inventory-II (BDI-II) at 12 Week Endpoint
Description: BDI-II is a 21-item patient-completed questionnaire designed to assess characteristics of depression. Each item is rated on a 4-point scale (0 = not present; 3 = present in the extreme). This questionnaire will be used to rate the severity of depressive symptoms and any improvement during the course of the trial. The total score ranges from 0 to 63; the higher the score, the more severe the depressive symptoms.
Time Frame: Baseline, 12 weeks
Population: Number of patients with a non-missing baseline and at least one post-baseline record.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 233 | 237
units on a scale | -5.53 (0.53) | -3.63 (0.52)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.007, ANCOVA — The p-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: BDI-II Total score change from baseline to endpoint = baseline BDI-II total score + treatment + pooled investigator; Least Squares Mean Difference = -1.89, 95% CI 2-sided [-3.25 to -0.53] — Least Squares Mean Difference = Duloxetine minus Placebo

5. Secondary Outcome: Change From Baseline in Clinical Global Impressions of Severity (CGI-S) at 12 Week Endpoint
Description: The Clinical Global Impressions of Severity (CGI-Severity) scale evaluates the severity of illness at the time of assessment. The score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline, 12 Weeks
Population: Number of patients with a non-missing baseline and at least one post-baseline record.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 231 | 237
units on a scale | -1.05 (0.07) | -0.71 (0.07)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — The p-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: CGI-S score change from baseline at endpoint = CGI-S score baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.34, 95% CI 2-sided [-0.51 to -0.16] — Least Squares Mean Difference = Duloxetine minus Placebo

6. Secondary Outcome: Change From Baseline in Beck Anxiety Inventory (BAI) at 12 Week Endpoint
Description: BAI is a 21-item patient-completed questionnaire designed to assess characteristics of anxiety. Each item is rated on a 4-point scale (0 = not present; 3 = present in the extreme). This questionnaire will be used to rate the severity of anxiety symptoms and any improvement during the course of the trial. The total score ranges from 0 to 63; the higher the score, the more severe the anxiety symptoms.
Time Frame: Baseline, 12 weeks
Population: Number of patients with a non-missing baseline and at least one post-baseline record.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 230 | 232
units on a scale | -3.14 (0.46) | -3.22 (0.46)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.907, ANCOVA — The p-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: BAI total score change from baseline to endpoint = baseline BAI total + treatment + pooled investigator; Least Squares Mean Difference = 0.07, 95% CI 2-sided [-1.13 to 1.27] — Least Squares Mean Difference = Duloxetine minus Placebo

7. Secondary Outcome: Change From Baseline in 36-Item Short-form Health Survey (SF-36) at 12 Weeks
Description: The patient-rated SF-36 consists of 36 questions covering eight health domains: physical functioning, bodily pain, role limitations due to physical problems, role limitations due to emotional problems, general health perceptions, mental health, social function, and vitality. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale, with higher scores indicating better health status or functioning. Two summary scores: the Physical Component Summary and the Mental Component Summary are constructed based on the eight SF-36 domains.
Time Frame: Baseline, 12 weeks
Population: Number of patients with a non-missing baseline and at least one post-baseline record.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 232 | 235
units on a scale
  Bodily Pain | 18.48 (1.33) | 13.26 (1.32)
  General Health | 9.33 (1.16) | 2.91 (1.15)
  Mental Health | 10.05 (1.17) | 2.61 (1.15)
  Physical Functioning | 13.52 (1.31) | 8.06 (1.30)
  Role-Emotional | 14.91 (2.57) | 5.13 (2.54)
  Role-Physical | 20.49 (2.51) | 18.90 (2.48)
  Social Functioning | 14.16 (1.52) | 7.49 (1.50)
  Vitality | 12.78 (1.34) | 8.47 (1.32)
  Physical Component Summary (PCS) | 5.96 (0.58) | 4.81 (0.57)
  Mental Component Summary (MCS) | 5.11 (0.69) | 1.28 (0.68)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value for Bodily Pain. The p-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: SF-36 subscale change from baseline at endpoint = SF-36 subscale at baseline + treatment + pooled investigator; Least Squares Mean Difference = 5.22, 95% CI 2-sided [1.76 to 8.67] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for General Health. The p-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: SF-36 subscale change from baseline at endpoint = SF-36 subscale at baseline + treatment + pooled investigator; Least Squares Mean Difference = 6.42, 95% CI 2-sided [3.41 to 9.43] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Mental Health. The p-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: SF-36 subscale change from baseline at endpoint = SF-36 subscale at baseline + treatment + pooled investigator; Least Squares Mean Difference = 7.44, 95% CI 2-sided [4.41 to 10.47] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value for Physical Functioning. The p-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: SF-36 subscale change from baseline at endpoint = SF-36 subscale at baseline + treatment + pooled investigator; Least Squares Mean Difference = 5.47, 95% CI 2-sided [2.06 to 8.88] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.004, ANCOVA — P-value for Role-Emotional. The p-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: SF-36 subscale change from baseline at endpoint = SF-36 subscale at baseline + treatment + pooled investigator; Least Squares Mean Difference = 9.78, 95% CI 2-sided [3.11 to 16.45] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.632, ANCOVA — P-value for Role-Physical. The p-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: SF-36 subscale change from baseline at endpoint = SF-36 subscale at baseline + treatment + pooled investigator; Least Squares Mean Difference = 1.59, 95% CI 2-sided [-4.93 to 8.11] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Social Functioning. The p-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: SF-36 subscale change from baseline at endpoint = SF-36 subscale at baseline + treatment + pooled investigator; Least Squares Mean Difference = 6.67, 95% CI 2-sided [2.73 to 10.61] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.015, ANCOVA — P-value for Vitality. The p-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: SF-36 subscale change from baseline at endpoint = SF-36 subscale at baseline + treatment + pooled investigator; Least Squares Mean Difference = 4.31, 95% CI 2-sided [0.84 to 7.79] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 9: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.134, ANCOVA — P-value for Physical Component Summary (PCS). The p-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: SF-36 subscale change from baseline at endpoint = SF-36 subscale at baseline + treatment + pooled investigator; Least Squares Mean Difference = 1.14, 95% CI 2-sided [-0.35 to 2.64] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 10: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Mental Component Summary (MCS). The p-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: SF-36 subscale change from baseline at endpoint = SF-36 subscale at baseline + treatment + pooled investigator; Least Squares Mean Difference = 3.83, 95% CI 2-sided [2.05 to 5.60] — Least Squares Mean Difference = Duloxetine minus Placebo

8. Secondary Outcome: Change From Baseline in Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (MGH-CPFQ) Total Score at 12 Week Endpoint
Description: The MGH-CPFQ is a self-report instrument consisting of seven questions pertaining to an individual's cognitive and physical well-being. Each question is rated 1 = "greater than normal" to 6 = "totally absent". Total score ranges from 7 to 42.
Time Frame: Baseline, 12 weeks
Population: Number of patients with a non-missing baseline and at least one post-baseline record.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 246 | 254
units on a scale | -4.88 (0.42) | -3.92 (0.41)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.083, ANCOVA — A priori threshold for statistical significance is 0.05; Model: MGH-CPFQ change from baseline at endpoint = MGH-CPFQ baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.96, 95% CI 2-sided [-2.05 to 0.13] — Least Squares Mean Difference = Duloxetine minus Placebo

9. Secondary Outcome: Change From Baseline in the Mood, Anxiety, Pain, Sleep, and Stiffness Likert Scale at 12 Week Endpoint
Description: Likert scales are patient-rated assessments. Mood: feeling low, sad or depressed; rated 0 = not feeling low, sad or depressed to 10 = feeling extremely low, sad or depressed. Anxious: anxious feelings; rated 0 = not feeling anxious to 10 = extremely anxious. Sleep: how much patient bothered by sleep difficulties; rated 0 = not bothered to 10 = extremely bothered. Pain: how much patient bothered by painful physical discomforts; rated 0 = not bothered to 10 = extremely bothered. Stiffness: how stiff patient felt in past 24 hours; rated 0 = not felt any stiffness to 10 = felt extremely stiff.
Time Frame: Baseline, 12 weeks
Population: Number of patients with a non-missing baseline and at least one post-baseline record.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 249 | 258
units on a scale
  Mood | -1.27 (0.17) | -0.52 (0.16)
  Anxiety | -1.22 (0.16) | -0.58 (0.16)
  Pain | -2.45 (0.18) | -1.73 (0.18)
  Sleep | -1.96 (0.19) | -1.47 (0.18)
  Stiffness | -2.54 (0.17) | -1.67 (0.17)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Mood. P-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: Likert scale change from baseline at endpoint = Likert scale baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.75, 95% CI 2-sided [-1.18 to -0.32] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value for Anxiety. P-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: Likert scale change from baseline at endpoint = Likert scale baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.64, 95% CI 2-sided [-1.05 to -0.22] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value for Pain. P-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: Likert scale change from baseline at endpoint = Likert scale baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.72, 95% CI 2-sided [-1.19 to -0.25] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.050, ANCOVA — P-value for Sleep. P-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: Likert scale change from baseline at endpoint = Likert scale baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.49, 95% CI 2-sided [-0.97 to -0.00] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Stiffness. P-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05; Model: Likert scale change from baseline at endpoint = Likert scale baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.87, 95% CI 2-sided [-1.32 to -0.43] — Least Squares Mean Difference = Duloxetine minus Placebo

10. Secondary Outcome: Number of Responders: 30% Improvement in Brief Pain Inventory Average Pain at 12 Week Endpoint
Description: Response was defined as at least 30% reduction from baseline to endpoint (last observation carried forward) for BPI average pain score. BPI average pain score assesses the severity of the average pain in the past 24 hours. The average severity score ranges from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: 12 Weeks
Population: Number of randomized patients with baseline and at least one post-baseline data.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 249 | 258
participants | 119 | 88
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.002, Fisher Exact — A priori threshold for statistical significance is 0.05

11. Secondary Outcome: Number of Responders: 50% Improvement in Brief Pain Inventory Average Pain Score at 12 Week Endpoint
Description: Response was defined as at least 50% reduction from baseline to endpoint (last observation carried forward) for BPI average pain score. BPI average pain score assesses the severity of the average pain in the past 24 hours. The average severity score ranges from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: 12 weeks
Population: Number of randomized patients with baseline and at least one post-baseline data.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 249 | 258
participants | 83 | 55
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.003, Fisher Exact — A priori threshold for statistical significance is 0.05

12. Secondary Outcome: Change From Baseline in Blood Pressure at 12 Week Endpoint
Time Frame: Baseline, 12 weeks
Population: Number of patients with a baseline and at least one post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 250 | 259
mm Hg
  Systolic Blood Pressure (SBP) | 1.09 (0.80) | -0.72 (0.78)
  Diastolic Blood Pressure (DBP) | 0.83 (0.51) | 0.31 (0.50)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.084, ANCOVA — P-value for Systolic Blood Pressure (SBP). A priori threshold for statistical significance is 0.05; Model: Change = baseline + treatment + pooled investigator; Least Squares Mean Difference = 1.82, 95% CI 2-sided [-0.25 to 3.88] — Least Squares Mean Difference = Duloxetine minus Placebo
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.434, ANCOVA — P-value for Diastolic Blood Pressure (DBP). A priori threshold for statistical significance is 0.05; Model: Change = baseline + treatment + pooled investigator; Least Squares Mean Difference = 0.52, 95% CI 2-sided [-0.79 to 1.84] — Least Squares Mean Difference = Duloxetine minus Placebo

13. Secondary Outcome: Change From Baseline in Heart Rate at 12 Week Endpoint
Time Frame: Baseline, 12 weeks
Population: Number of patients with a baseline and at least one post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 250 | 259
beats per minute (bpm) | 1.76 (0.50) | -0.20 (0.49)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA — A priori threshold for statistical significance is 0.05; Model: Change = baseline + treatment + pooled investigator; Least Squares Mean Difference = 1.96, 95% CI 2-sided [0.67 to 3.26] — Least Squares Mean Difference = Duloxetine minus Placebo

14. Secondary Outcome: Number of Patients With Columbia Suicide Severity Rating Scale (CSSR-S) Events (Behaviors, Ideations, Acts)
Description: C-SSRS: scale capturing occurrence, severity, and frequency of suicide-related thoughts and behaviors. Number of patients with suicidal behaviors, ideations, and acts are provided. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation: a "yes" answer to any one of 5 suicidal ideation questions, which includes wish to be dead, and 4 different categories of active suicidal ideation. Suicidal act: a "yes" answer to actual attempt or completed suicide.
Time Frame: Baseline through 12 Weeks
Population: Number of randomized patients.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 263 | 267
participants
  Suicidal Ideation | 6 | 7
  Suicidal Behavior | 0 | 0
  Suicidal Acts | 0 | 0
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact — P-value for Suicidal Ideation. A priori threshold for statistical significance is 0.05

15. Secondary Outcome: Change From Baseline in Weight at 12 Week Endpoint
Time Frame: Baseline, 12 weeks
Population: Number of patients with a baseline and at least one post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 249 | 259
kilograms (kg) | -0.62 (0.15) | 0.21 (0.14)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — A priori threshold for statistical significance is 0.05; Model: Change = baseline + treatment + pooled investigator; Least Squares Mean Difference = -0.83, 95% CI 2-sided [-1.21 to -0.45] — Least Squares Mean Difference = Duloxetine minus Placebo

ADVERSE EVENTS:
Time Frame: These are the adverse events which occurred during the 12 week acute double-blind phase.
Arm/Group | Duloxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/263 | 6/267
Other Adverse Events (participants affected / at risk) | 217/263 | 189/267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=263) | Placebo (N=267)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=263) | Placebo (N=267)
Constipation (Gastrointestinal disorders) | 35 (35) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 27 (30) | 12 (12)
Dry mouth (Gastrointestinal disorders) | 31 (31) | 12 (12)
Nausea (Gastrointestinal disorders) | 83 (87) | 26 (28)
Vomiting (Gastrointestinal disorders) | 12 (15) | 2 (2)
Fatigue (General disorders) | 25 (26) | 19 (19)
Upper respiratory tract infection (Infections and infestations) | 13 (13) | 13 (14)
Decreased appetite (Metabolism and nutrition disorders) | 13 (13) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 11 (15)
Dizziness (Nervous system disorders) | 26 (27) | 14 (15)
Headache (Nervous system disorders) | 45 (48) | 24 (28)
Somnolence (Nervous system disorders) | 15 (16) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 11 (11)
Insomnia (Psychiatric disorders) | 24 (27) | 19 (20)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 23 (24) | 4 (4)
Hot flush (Vascular disorders) | 13 (14) | 2 (2)
Irritability (General disorders) | 3 (3) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days